CLINICAL TRIAL: NCT05901701
Title: Effect of Low-Level Laser Therapy Versus CAD/CAM Michigan Splint on Patients With Temporomandibular Muscle Disorders Randomized Clinical Trial
Brief Title: Efficacy of Low Level LASER Therapy in Treating Temporomandibular Muscle Disorders
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IR112207
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2022-11

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Low level LASER therapy; Michigan splint; Electromyogram; Myofascial pain
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Group A: Patients received applications of low-level laser therapy. Group B: Patients received hard occlusal splints (Michigan splints).
Who Masked: Outcomes Assessor
Masking Description: Blocked randomization technique was used to divide the patients into two equal groups using sealed envelopes, the person who was in charge for randomization was blinded to the group allocation of the patients. The outcome assessor also didn't know the allocated groups, and the patients were instructed not to mention their groups to the assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LASER group (Experimental): Group A: Patients received applications of low-level laser therapy using semiconductor InGaAsp diode LASER type 940 nm with continuous mode of operation, with time of application 180 sec per session for 12 sessions.
  Interventions: Radiation: Low Level LASER therapy
- Splint group (Active Comparator): Group B: Patients received hard occlusal splints (Michigan splints), used for 3 months during sleeping then the patient stops using it and told to only wear it if discomfort return usually during stressful times.
  Interventions: Device: Hard occlusal splint

INTERVENTIONS:
Radiation: Low Level LASER therapy — using semiconductor InGaAsp diode LASER type 940 nm with continuous mode of operation, with time of application 180 sec per session for 12 sessions.
  Arms: LASER group
Device: Hard occlusal splint — 2 mm thickness occlusal splint constructed over the maxillary arch using CAD/CAM technology.
  Other Names: Michigan splint
  Arms: Splint group

SUMMARY:
This study aimed to evaluate the sustainability of the efficacy of using low level laser therapy and CAD/CAM Michigan splint in improving the range of mandibular movements, muscle activity and reducing the pain.

DETAILED DESCRIPTION:
56 female patients were randomly divided into two groups, Group A: Patients received applications of low-level laser therapy using semiconductor InGaAsp diode LASER type 940 nm with continuous mode of operation, with time of application 180 sec per session for 12 sessions. Group B: Patients received hard occlusal splints (Michigan splints) of 2 mm thickness constructed on their upper teeth, the hard occlusal splint was 3D digitally printed. ARCUS digma facebow was used to evaluate the range of mandibular movements affected from TMJ problems. The opening measurements of the patient were taken using a millimeter ruler. Electromyogram (EMG) was used to evaluate muscle activity. Visual analogue scale (VAS) was used to evaluate the pain intensity. All was done before the beginning of the treatment at three and six months follow up period.

ELIGIBILITY:
Inclusion Criteria: tenderness in the TMJ or muscles of mastication (e.g., temporalis and masseter) that might get worse in the morning or with eating, headache, periauricular pain, teeth wear that appears in the form of multiple smooth shinny facets, teeth mobility, and malocclusion

Exclusion Criteria:

* pregnant females, breast feeders, patients having pacemakers, heart disease, tumors, general connective tissue disease e.g., Rheumatoid arthritis, psychiatric disorders, skeletal morphology as class II or III, TMJ clicking sounds, local skin infection over the masseter or temporalis, symptoms that may be referred to other disorders of orofacial region (tooth ache, trigeminal neuralgia, migraine), or patients using medications such as Muscle relaxant, Steroids, Dopamine precursors like L dopa and Aminoglycoside
* Vulnerable groups (prisoners, mental disorders, patients not capable of decision making).

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Electromyographic muscle activity | Measured 3 times through 6 months from the beginning of the treatment. (0,3,6 months)
  The change in muscle activity was assessed using EMG in terms of Microvolt
Range of mandibular movement | Measured 3 times through 6 months from the beginning of the treatment. (0,3,6 months)
  The increase in the range of movement measured using ARCUS digma in terms of angular inclination.

SECONDARY OUTCOMES:
Pain intensity | Measured 3 times through 6 months from the beginning of the treatment. (0,3,6 months)
  The degree of pain is assessed using a 10 cm scale (VAS)
Mouth opening | Measured 3 times through 6 months from the beginning of the treatment. (0,3,6 months)
  degree of mouth opening in cm using ruler

CONTACTS AND LOCATIONS:
Overall Officials: Rami M Ghali, professor, Study Director — oral and maxillofacial prosthodontics department, faculty of dentistry, Ain Shams University; Amany M Farahat, PhD, Principal Investigator — Oral and Maxillofacial prosthodontics department, faculty of dentistry, Ain Shams University; Dina E Bahig, PhD, Principal Investigator — Oral and Maxillofacial prosthodontics department, faculty of dentistry, Ain Shams University
Locations (1):
- faculty of dentistry, Ain Shams University, Cairo, Egypt